CLINICAL TRIAL: NCT01917032
Title: Effect of Home-fortification With Micronutrient Powder Sprinkles in Hematologic and Nutritional Status in Preschool Children in Medellín: a Randomized Clinical Trial.
Brief Title: Effect of Home-fortification With Sprinkles in Hematologic and Nutritional Status in Preschool Children in Medellín
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Cristian Vargas G. MD, Student, CES University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPRINK001
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Malnutrition
Keywords: Trace Elements; Preschool; Malnutrition; Fortified Food
MeSH Terms: conditions — Malnutrition | interventions — Iron; Zinc; Folic Acid; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sprinkles (Active Comparator): Micronutrient Powder Sprinkles 1 gram orally on weekdays during 11 weeks
  Interventions: Dietary Supplement: Sachets containing a blend of micronutrients in powder form (Iron, Zinc, Folic Acid, Vitamin A and C), sprinkled onto home made food
- Placebo (Placebo Comparator): Maltodextrin 1 gram orally on weekdays during 11 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Sachets containing a blend of micronutrients in powder form (Iron, Zinc, Folic Acid, Vitamin A and C), sprinkled onto home made food — 1 g orally on weekdays during 11 weeks
  Other Names: Chispitas; Sprinkles
  Arms: Sprinkles
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
Objective: To acquire the local scientific evidence, to evaluate the effects of micronutrient Sprinkles™ powder, both the nutritional status and haematological values in the vulnerable preschool population, to corroborate the reported benefits of the experiences in other countries.

Question: Will it improve the nutritional status and hematological levels after the home fortification with Sprinkles in children of two child care centres in the city of Medellin, in 2013?

Hypothesis: At the end of intervention, hematologic levels and anthropometric indicators will be better in the intervention group with Sprinkles, compared with the placebo group.

Design: Randomized clinical trial, triple-blind and placebo-controlled.

Participants: Two groups of 50 children each, aged between 5 and 59 months, not anemic or with severe malnourished, full-time assistants to two children's centres that have the same alimentation menu.

Intervention: The daily diet will be supplemented with sprinkles in one of the children's centres and will be compared anthropometric and hematological values before and after with a group receiving the same diet with placebo.

Outcome measures: Nutritional status (anthropometric measures) and haematological values (hemoglobin, ferritin, transferrin and folate).

ELIGIBILITY:
Inclusion Criteria:

* Assistance to children's centres full day (8 hours).
* Age 5 to 59 months.

Exclusion Criteria:

* Anemia (hemoglobin less than 11 g / dl).
* Current supplementation with a product formulated by a health professional as a part of a nutritional recovery.
* Denial for informed consent signing by parents or legal guardians.
* Diagnosis of severe acute malnutrition by anthropometric measurements.

Ages: 5 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 10 weeks
  Hemoglobin quantitation for laboratory tests (g/dl)

SECONDARY OUTCOMES:
Transferrin | 10 weeks
  Transferrin quantitation for laboratory tests (mg/dl)

OTHER OUTCOMES:
Child Growth Indicators | 10 weeks
  Anthropometric measurements as indicators of child growth and nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Vargas, MD, Principal Investigator — CES University; Juliana Orozco, Nutricionist, Principal Investigator — CES University; Juliana Sánchez, Dentist, Study Chair — CES University; Liliana Montoya, Epidemiology, Study Director — CES University; Javier Chica, Veterinarian, Study Chair — CES University; Maylen Rojas, Epidemiology, Study Chair — CES University; Óscar Villada, MD, Study Chair — CES University; Alejandro Díaz, Pediatrist, Study Chair — CES University
Locations (1):
- Fundación de Atención a la Niñez (FAN), Medellín, Ant, Colombia